CLINICAL TRIAL: NCT05200234
Title: Improving Cerebral Blood Flow and Cognitive Function in Patients With Asymptomatic Intracranial / Carotid Stenosis With Nattokinase (ICC-PACS): a Randomized Controlled Trial
Brief Title: Improving Cerebral Blood Flow and Cognitive Function in Patients With Asymptomatic Intracranial / Carotid Stenosis With Nattokinase (ICC-PACS)
Acronym: ICC-PACS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ICC-PACS
Record Dates: First submitted 2022-01-17; First posted 2022-01-20 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Cerebral Blood Flow; Cognitive Function
Keywords: Intracranial / Carotid Stenosis; Cerebral Blood Flow; Cognitive Function
MeSH Terms: conditions — Carotid Stenosis | interventions — nattokinase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Nattokinase + standard medical treatment
  Interventions: Drug: Nattokinase
- Control group (Placebo Comparator): Placebo + Standard medical treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nattokinase — Nattokinase + standard treatment
  Arms: Intervention group
Drug: Placebo — Placebo+ standard treatment
  Arms: Control group

SUMMARY:
A randomized controlled trial will be conducted. Patients with asymptomatic intracranial / carotid stenosis will be randomized into two arms (1:1): an intervention arm and a control arm. Patients in the intervention arm will be treated with standard medical treatment combined with Natto Products V, whereas Patient in the control arm will be treated with only standard medical treatment . And the impact of Natto Products V on improving cerebral blood flow and cognitive function in patients with asymptomatic intracranial / carotid stenosis will be assessed by neuropsychological scale and multimode magnetic resonance imaging.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 40 years
* ≥ 50% stenosis in unilateral intracranial / carotid artery
* Written informed consent available

Exclusion Criteria:

* Previous history of major head trauma and any intracranial surgery
* Intracranial abnormalities, such as intracerebral hemorrhage, subarachnoid hemorrhage and other space occupying lesions
* Extrapyramidal symptoms or mental illness which may affect neuropsychological measurement
* severe loss of vision, hearing, or communicative ability
* plan to be treated with surgery

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-01-13 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in the scores of Montreal Cognitive Assessment | 6 months
  Total score of 30

SECONDARY OUTCOMES:
Changes in the scores of Mini-mental State Examination | 6 months
  Total score of 30
Changes in cerebral blood flow in the territory of the culprit artery | 6 months
Changes in the scores of Colour Trail Test | 6 months
Changes in the scores of Hopkins Verbal Learning Test | 6 months
Changes in the scores of clock drawing test | 6 months
Changes in the scores of Animal Fluency Test | 6 months
Changes in the scores of Olfactory stick test | 6 months
Incidence of stroke event including ischemic and hemorrhagic stroke | 6 months
Changes in cerebral glymphatic function | 6 months
  assessed by non-invasive diffusion tensor image analysis along the perivascular space (ALPS-index)
Changes in metabonomics | 6 months
  include blood and fecal samples

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affilated Hospital of Zhejiang University, School of Medicine, Hangzhou, Zhejiang, China